CLINICAL TRIAL: NCT05403619
Title: Impact of an Enhanced Focused Cardiac Ultrasound on Treatment Modifications in a Population of Internal Medicine Patients: Retrospective Study
Brief Title: Enhanced FoCUS in Patients With Shortness of Breath
Acronym: eFOCUS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: eFOCUS 1
Record Dates: First submitted 2022-05-19; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Shortness of Breath; Acute Respiratory Failure
Keywords: Acute decompensated heart failure; Pneumonia; Pulmonary Embolism; Ultrasound
MeSH Terms: conditions — Dyspnea; Pneumonia; Pulmonary Embolism | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients hospitalized for shortness of breath with realization of an enhanced FoCUS
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Cardiac Ultrasound in order to explore the causes of shortness of breath
  Other Names: Focused cardiac Ultrasound

SUMMARY:
Retrospective observational study performed in a internal medicine ward of a French university hospital. Included patients were hospitalized for acute shortness of breath who have benefited from a eFOCUS which was defined as a focused cardiac Ultrasound with utilization of Doppler measurements.

The objectives were the therapeutic and diagnosis changes induced by eFoCUS. The primary endpoint was defined by the pooled introduction or discontinuation of diuretics, antibiotics or anticoagulants associated with eFoCUS results.

DETAILED DESCRIPTION:
It was a retrospective observational study performed in a internal medicine ward of a French University Hospital. Patients were identified in the hospital database, pertinent features and eFoCUS findings were extracted and anonymized.

Inclusion criteria:

* Adult patients admitted to an internal medicine ward from the ED for acute shortness of breath.
* Realization of an eFoCUS prescribed by the physician in charge of the patient

Exclusion criteria:

• Comprehensive echocardiography already performed Methods For each identified patient, pertinent data (demography, initial diagnosis and treatment (diuretics, antibiotics, anticoagulants)) and eFoCUS findings were extracted from the hospital files, anonymized and entered in a LibreOffice spreadsheet. Extracted diagnosis were gathered into the following categories: Community-acquired pneumonia (CAP), Acute cardiogenic pulmonary edema (ACPE), Pulmonary embolism (PE), Chronic Obstructive Pulmonary Disease (COPD) and other (OTHER).

Objectives and endpoints

* The main objective was the therapeutic change induced by eFoCUS. The primary endpoint was defined by the pooled introduction or discontinuation of diuretics, antibiotics or anticoagulants associated with eFoCUS results.
* The secondary objectives were diagnosis modifications induced by eFoCUS. Data analysis
* Numerical data were presented as mean ± SD or as median with interquartile range depending on the normality. The paired Student's t-test was used to compare normally distributed data. The chi-square test was used for the comparison of noncontinuous variables expressed as proportions. A p-value <0.05 was considered significant. All p-values were two-sided. Statistical analysis was realized with R (4.03.3) in the Rstudio® environment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to a internal medicine ward from the ED for acute shortness of breath.
* Realization of an eFoCUS prescribed by the physician in charge of the patient

Exclusion Criteria:

* Comprehensive echocardiography already performed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acute shortness of breath
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Pooled introduction or discontinuation of diuretics, antibiotics or anticoagulants | up to 24 hours after eFoCUS
  Number of patients for whom there was an introduction or discontinuation of diuretics, antibiotics or anticoagulants associated with Focused cardiac ultrasound

SECONDARY OUTCOMES:
Changes of diagnostic categories associated with eFOCUS | up to 24 hours after eFoCUS
  Number of patients for whom the diagnostic category (pneumonia, acute cardiac failure, pulmonary embolism, COPD, other) was modified after Focused cardiac ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No